CLINICAL TRIAL: NCT03155906
Title: Integrated Treatment of Hepatitis C Virus Infection Among Patients With Injecting Drug Abuse:a Randomised Controlled Trial (INTRO-HCV)
Brief Title: Integrated Treatment of Hepatitis C Virus Infection
Acronym: INTRO-HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); Forskningsrådet (Unknown); Helse Vest (Other); University of Bergen (Other); Folkehelseinstituttet (Unknown); Bergen kommune (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2017/51/REK vest
Record Dates: First submitted 2017-05-04; First posted 2017-05-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C, Chronic; Opioid Dependence, on Agonist Therapy
Keywords: Chronic hepatitis C; Opiate Substitution Treatment; Integrated Delivery of Health Care; Substance Abuse Treatment Centers
MeSH Terms: conditions — Hepatitis C, Chronic; Opioid-Related Disorders | interventions — Delivery of Health Care; Delivery of Health Care, Integrated

STUDY DESIGN:
Intervention Model Description: A multicentre, randomised controlled clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Even though complete blinding is regarded as difficult, there will be some degree of blinding/masking. Randomisation will be disclosed to physician and other health care staff providing OST treatment, but not to research nurses conducting data collection for outcomes. Patients will be informed of the follow-up they will receive, but not on other follow-up alternatives that are used or the exact hypotheses for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated treatment (Experimental): Patients randomised to receive integrated treatment will be counselled on treatment by physician working at MAR outpatient clinic where patient receive OST care, and will receive medication and follow-up at the same MAR outpatient clinic. Treatment medication will be given in line with national guidelines with a close and integrated follow-up.
  Interventions: Other: Health care delivery
- Standard treatment (Active Comparator): Those randomised to receive standard treatment will be offered referral for standard HCV treatment at a medical ward hospital clinic. Treatment medication will be given in line with national guidelines.
  Interventions: Other: Health care delivery

INTERVENTIONS:
Other: Health care delivery — Integrated HCV treatment within the OST clinics will compared to standard treatment. Those who are eligible to receiving treatment in line with national guidelines, have no exclusion criteria and consent to study participation, will be randomised to either standard or integrated treatment. For the integrated treatment, treatment initiation, follow-up and delivery of medication will be given at a MAR outpatient clinic where they already receive care including OST. Those randomised to standard treatment will be referred to a medical ward clinic for assessment of treatment initiation and follow-up. Assessment of outcomes will be done 12 weeks after completed treatment and adherence will be assessed at 4, 8 and 12 weeks after initiation of treatment.
  Other Names: Integrated health care

SUMMARY:
INTRO-HCV is a multicentre randomised controlled clinical trial that will compare the efficacy of integrated treatment of chronic hepatitis C virus infection (HCV) within medically assisted rehabilitation (MAR) clinics providing opioid substitution therapy (OST) compared to standard treatment. The trial will recruit approximately 250 HCV infected in Bergen and Stavanger and about 1000 in a linked observational study.

Intervention: Integrating diagnostic and treatment follow-up for HCV treatment into MAR outpatient clinics in Bergen and Stavanger including testing for HCV, counselling and treatment evaluation and treatment delivery.

Primary objectives: Compare the effect of integrated HCV treatment assessed with sustained virological response at 12 weeks between the MAR outpatient clinics in Bergen and Stavanger (intervention arm) with standard treatment provided after referral to infectious disease clinics among patients who receive OST having HCV Secondary objectives: Compare treatment adherence between the intervention and control arms, and assess changes in quality of life, fatigue and psychological well-being before and after HCV treatment, as well as changes in drug use, infection related risk behavior, and risk of reinfection among those with sustained virological response.

Main endpoint: Sustained virological response of HCV at 12 weeks (± 10 days) Study population: The target group will be patients receiving care with MAR from involved outpatient clinics in Bergen, Sandnes and Stavanger who are chronically infected with HCV and eligible for treatment according to national guidelines.

Study duration: Participants will be included and followed up at least annually for the total study duration between 2017 and 2021.

Expected outcome: This study will inform on the relative advantages and disadvantages of an integrated treatment program for HCV into MAR compared to standard care aiming to increase access to treatment and improved treatment adherence. If the integrated treatment structure is found to be safe and efficacious, it can be considered for further scale-up.

DETAILED DESCRIPTION:
Rationale Globally, about 71 million people are chronically infected with chronic hepatitis C virus infection (HCV) and approximately 700,000 are dying annually of related complications. It has been estimated to be 10-20,000 people in Norway have chronic HCV. People who inject drugs represent around 75% of these, most being infected with HCV through sharing of syringes and other user equipment. HCV and hepatitis B are both among the leading causes to liver disease and transplantation worldwide. Prevention and control has to date unfortunately shown to be difficult.

Among people with opioid addiction and HCV, a third develops severe complications within three decades. Within the same group and after 50 years of age, liver disease is as common as risk of death as overdose. Reports from medically assisted rehabilitation (MAR) clinics delivering opioid substitution therapy (OST) in Norway indicate that more than half of the patients receiving OST have a HCV. Chronic HCV substantially increases the risk of severe complications such as liver failure and death within two to three decades. The mean age of OST patients in Norway is 42 years and is currently increasing, and a large group have had HCV for more than twenty years. Reaching these patients with treatment is of critical importance to avoid deaths and reduced quality of life, as well as preventing large costs related to future treatment of end stage liver disease. Treatment for HCV has been available for several decades, and weekly injections with interferon in combination with daily ribavirin tablets for 16 to 48 weeks has until recently been the standard treatment. These medications have been shown to give frequent and to some degree serious side effects, with around 40% not achieving sustained virological response (SVR). These aspects combined with a fear among many clinicians of reinfection among those being treated and an expectation of poor treatment adherence in this group, has probably been the reasons for few patients having been treated yet. However, studies assessing treatment adherence indicate good adherence among patients receiving OST. Even if around 6% of those who are successfully treated among people who inject drugs are reinfected annually, treatment is not only important for those who are treated, but will also contribute to reduce the HCV infectious burden and the risk of spread within the population.

During the last years, development of new highly effective tablet-based direct acting antiretroviral medications, usually being curative within 8 to 16 weeks, has radically changed the HCV treatment. These treatments have less side effects than those used earlier and give opportunities to cure most of the HCV infected. Even if they are expensive, British assessments indicate that they are cost effective as universal coverage with antiretroviral treatment could prevent large expenses related to future complications. Thus, the Norwegian Medicines Agency approved many of these new antiretroviral treatments in 2014. Nevertheless, a recent Norwegian study indicated that only 14% of OST patients with chronic HCV had received HCV treatment. Currently, the high burden of HCV among people who inject drugs is among the largest challenges within the MAR field, within a group that is also underrepresented in clinical research.

Patients with drug addiction have a high disease burden, generally have more difficulties in obtaining adequate health care compared with the general population, on top of knowledge gaps in terms of health status and how to deliver proper treatment and follow-up. This is particularly the case among people who inject drugs.

There is a need for new approaches to reach more of those in need of treatment while ensuring high-quality care. To reach patients with drug addiction, it seems to be necessary to use a model of health care focusing on interdisciplinarity, accessibility, close and frequent follow-ups.

Department of Addiction Medicine at Haukeland University Hospital in Bergen and OST in Stavanger have adopted an integrated treatment and care model for patients receiving OST with follow-up by physicians, nurses, social workers and psychologists on nearly a daily basis with observed intake of the OST medications. This model for treatment of OST patients is unique for Bergen and Stavanger, also in an international perspective. This makes it an excellent platform to test out integration of HCV treatment aiming to improve health and life span of a vulnerable group, and at the same time gathering knowledge which traditionally has been difficult to obtain.

This research project designed as a randomised controlled trial done in parallel with an observational study will test whether integrated treatment of HCV linked to the MAR outpatient clinics to patients with chronic HCV will have better outcomes in terms of reduction in HCV.

The main aim of the study is to:

1. Compare the effect of integrated HCV treatment between the OST outpatient clinics in Bergen and Stavanger (intervention arm) with standard treatment provided after referral to infectious disease clinics among patients who receive OST having HCV

Primary objectives

* Compare the proportion with sustained virological response of HCV at 12 (10 - 14) weeks between those randomised to intervention and control arms
* Compare the proportion initiating treatment (taking at least one tablet or collecting prescription from pharmacy) between the intervention and control arms

Secondary objectives

* Assessing the incidence and prevalence of HCV at the OST outpatient clinics in Bergen, Stavanger, Sandnes, and at municipal primary health care clinics
* Compare treatment adherence between the intervention and control arms
* Assess the risk of reinfection among those with sustained virological response and compare between the arms
* Assess changes in quality of life, fatigue and psychological well-being before and after HCV treatment
* Assess changes in drug use and infection related risk behaviour before and after HCV treatment
* Estimate incidence and prevalence of HCV infection among people who inject drugs in Bergen, Stavanger and Sandnes being followed up at OST outpatient clinics or people who inject drugs followed up at primary health care clinics
* Estimate incidence and prevalence of HCV infection among people who inject drugs in Bergen, Stavanger and Sandnes being followed up at OST outpatient clinics or people who inject drugs followed up at primary health care clinics.

Study design and methodology Hypothesis Our hypothesis is that a model with integrated treatment of HCV linked to the OST outpatient clinics to patients with chronic HCV will have better outcomes in terms of reduction in HCV (sustained virological response) compared to the current model where patients are referred to a hospital outpatient clinic.

General outline:

The investigators will conduct a multicentre randomised controlled clinical trial without pharmaceutical industry involvement assessing integrated HCV treatment within the MAR clinics compared to standard treatment. The research project will be closely integrated with clinical care, and the research activities are planned during a planned scale-up of HCV treatment.

Department of Addiction Medicine at Haukeland University Hospital in Bergen and MAR in Stavanger have adopted an integrated treatment and care model for patients receiving OST. In Bergen, MAR outpatient clinics have been established in each district where the patients are followed up by health and social workers on nearly a daily basis with observed intake of the OST medications. Every month, the MAR clinics have a total of 6,000 patient visits among the approximately 500 patients. This group of patients have a large morbidity burden and have to limited degree been able to access other standard health care. Each of the MAR outpatient clinics is staffed by a consultant and a physician specialising in addiction medicine in addition to nurses, social workers, and several of the clinics also being staffed by a psychologist. The remaining 550 OST patients in Bergen are followed up mainly in primary care clinics. A close collaboration has been established between the Department of Addiction Medicine and the Agency for addiction and mental health in Bergen municipality, who is responsible for the care in several of the primary health clinics in Bergen. This model for treatment of MAR patients is unique for Bergen, also in an international perspective. MAR Stavanger has a relatively similar structure. MAR Stavanger is responsible for the MAR treatment of approximately 460 patients within their area. Of these, 120 patients are linked to the MAR outpatient clinic in the centre of Stavanger and 70 are linked to a similar clinic in Sandnes. The treatment model in Bergen and Stavanger is an excellent platform to test out integration of HCV treatment aiming to improve health and life span of a vulnerable group, and at the same time gathering knowledge which traditionally have been very difficult to obtain.

All patients will be assessed for HCV including genotyping among those who test HCV RNA positive. Those who are eligible to receiving treatment in line with national guidelines, have no exclusion criteria and consent to study participation, will be randomised to either standard or integrated treatment. In standard treatment, follow-up and treatment will be given at hospital clinics. For the integrated treatment, treatment will be given at a MAR outpatient clinic where they already receive care including MAR. Assessment of outcomes will be done 12 weeks after completed treatment and adherence will be assessed at 4, 8 and 12 weeks after initiation of treatment.

Main study outcomes

1. Sustained virological response of HCV at 12 (10 - 14) weeks after completed treatment
2. Treatment initiation

Milestones and duration of the study The duration of the study will be five years. Ethical clearance and complete protocol will be completed within the first half of 2017. Planned initiation of data collection is May 2017 with gradual scaling up of data collection throughout 2017. Recruitment will continue throughout 2019 and further follow-up throughout 2021. Analyses and reporting will be initiated from mid of 2018 for some of the observational studies while assessment of the trial will be conducted when at least 200 patients have completed follow-up at 12 weeks after end of treatment.

Study population and setting In Bergen, there are MAR policlinics in each district. Around half of the patients have frequent contact with the outpatient clinic several times per week. A substantial proportion receive OST-medications at a local pharmacy or through their general practitioner. In addition a few receive OST-medications at the aftercare centre Albatrossen, in schools or prisons. Most outpatient clinics are staffed with physicians (including both non-specialists or linked consultants/specialists), psychologists, and nurses or social workers/educators. In addition, a decentralised unit has 228 patients in 18 municipalities, where most patients receive OST from a local pharmacy or through their general practitioner (GP). For more information, see https://helse-bergen.no/avdelinger/rusmedisin/rusmedisin-lar In addition, there are several patients receiving care without MAR at the municipal care centres at Wergeland, Nesttun og Gyldenpris (Strax-huset). For further description of these, see https://www.bergen.kommune.no/aktuelt/tema/tiltak-mot-rus/article-109220.

LAR Stavanger has one more centralised outpatient clinic in Stavanger and a smaller clinic in the nearby city Sandnes.

The research project will improve understanding on how the structure of health care impacts on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Receiving OST from included outpatient clinic
* Chronically infected with HCV (HCV RNA positive and also HCV RNA positive or anti-HCV at least 6 months before inclusion)
* Eligible for treatment according to national guidelines (criteria specified below)
* Obtaining informed consent

At the time of study initiation , eligibility for treatment according to national guidelines was defined as follows:

* Genotype 1 and 4 independent of degree of fibrosis
* Genotype 2 and 3, dependent on significant fibrosis.

Significant fibrosis will be assessed with FibroScan indicating elastography of above 7 kPa. Where elastography cannot be obtained, significant fibrosis will be assessed with AST to platelet ratio index (APRI score) of > 0.7 (http://www.hepatitisc.uw.edu/page/clinical-calculators/apri), i.e.

APRI = ASAT levels (in IU/L) / 40 (upper normal levels of ASAT in IU/L) / platelet count (109/L). An APRI score greater than 0.7 had a sensitivity of 77% and specificity of 72% for predicting significant hepatic fibrosis.

Exclusion Criteria:

* Co-infection with HIV
* Severe extrahepatic HCV associated diseases (e.g. cerebral vasculitis, cryoglobulinemia/membranoprolifereative glomerulonephritis (MPGN), renal failure (eGFR <30), polyarthritis)
* Decompensated liver failure assessed with Child-Pugh (CP) score (>6 points, class B and C)
* Currently receiving treatment for HCV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Sustained virological response of HCV at 12 | At 12 (10 - 14) weeks after completed treatment
  Sustained virological response of HCV will be assessed by HCV RNA at 12 (range 10 - 14) weeks after completed treatment
Treatment initiation | 6 months after diagnosing HCV in need of treatment
  Treatment initiation within 6 months after diagnosing HCV in need of treatment (in line with national guidelines). This will be assessed through observation in intervention and in reported obtainment from pharmacies of the prescribed drugs

SECONDARY OUTCOMES:
Treatment adherence | At 4, 8 (and 12 for treatment recommended beyond 8 weeks) weeks after treatment initiation
  Treatment adherence will be assessed by proportion of doses observed being taken in intervention group and reported obtainment from pharmacies of the prescribed drugs combined with self-reported questions on adherence collected at 4, 8 (and 12 for treatment recommended beyond 8 weeks) weeks after treatment initiation. The self-reported question categorises adherence during last four weeks into rarely, sometimes but less than half of the doses, between 50 and 80% of the doses, more than 80% of the doses, and always (95% of doses or more)
Changes in quality of life | At 12 weeks after treatment compared to before treatment
  Changes in quality of life will be assessed with EQ-5D-5L at 12 weeks after treatment compared to before treatment
Changes in fatigue | At 12 weeks after treatment compared to before treatment
  Changes in fatigue will be assessed with the Fatigue Symptom Scale (FSS) at 12 weeks after treatment compared to before treatment
Changes in psychological well-being | At 12 weeks after treatment compared to before treatment
  Changes in psychological well-being will be assessed with the Norwegian validated translation ten time version of Hopkins Symptom Checklist (SCL-10) at 12 weeks after treatment compared to before treatment
Changes in drug use | At 12 weeks after treatment compared to before treatment
  Assessment of changes in drug use will be assessed with self-reported use of the following drug categories the last 30 days, the last 12 months and ever: Alcohol, tobacco, cannabis, amphetamines, cocaine, heroin, other opioids not prescribed by physician, benzodiazepines or z-hypnotics, hallusinogens, solvents and gamma hydroxybutyrate (GHB), anabole steroids and other drugs at 12 weeks after treatment compared to before treatment
Changes in drug infection related risk behaviour | At 12 weeks after treatment compared to before treatment
  Assessment of changes in infection related risk behaviour will be assessed with questions assessing sharing of needles and other user equipment before and after HCV treatment at 12 weeks after treatment compared to before treatment
Changes in incidence of HCV | Assessed annually at follow-up assessments, up to 3 years
  Changes in incidence of HCV at the OST outpatient clinics in Bergen, Stavanger, Sandnes during the follow-up periode (2017-2019). Re-infections will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Lars T Fadnes, MD, PhD, Principal Investigator — Department of Addiction Medicine, Haukeland University Hospital; Else-Marie Løberg, MA, PhD, Study Chair — Department of Addiction Medicine, Haukeland University Hospital
Locations (2):
- Norway (2):
  - Department of Addiction Medicine, Haukeland University Hospital, Bergen, Hordaland
  - LAR Helse Stavanger HF, Stavanger, Rogaland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohd Hanafiah K, Groeger J, Flaxman AD, Wiersma ST. Global epidemiology of hepatitis C virus infection: new estimates of age-specific antibody to HCV seroprevalence. Hepatology. 2013 Apr;57(4):1333-42. doi: 10.1002/hep.26141. Epub 2013 Feb 4. PMID 23172780
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Background] Dalgard O, Jeansson S, Skaug K, Raknerud N, Bell H. Hepatitis C in the general adult population of Oslo: prevalence and clinical spectrum. Scand J Gastroenterol. 2003 Aug;38(8):864-70. doi: 10.1080/00365520310004542. PMID 12940441
- [Background] Kielland KB, Delaveris GJ, Rogde S, Eide TJ, Amundsen EJ, Dalgard O. Liver fibrosis progression at autopsy in injecting drug users infected by hepatitis C: a longitudinal long-term cohort study. J Hepatol. 2014 Feb;60(2):260-6. doi: 10.1016/j.jhep.2013.09.022. Epub 2013 Oct 2. PMID 24096048
- [Background] Kielland KB, Skaug K, Amundsen EJ, Dalgard O. All-cause and liver-related mortality in hepatitis C infected drug users followed for 33 years: a controlled study. J Hepatol. 2013 Jan;58(1):31-7. doi: 10.1016/j.jhep.2012.08.024. Epub 2012 Sep 4. PMID 22960427
- [Background] Seeff LB. Natural history of chronic hepatitis C. Hepatology. 2002 Nov;36(5 Suppl 1):S35-46. doi: 10.1053/jhep.2002.36806. PMID 12407575
- [Background] Hajarizadeh B, Grebely J, Dore GJ. Epidemiology and natural history of HCV infection. Nat Rev Gastroenterol Hepatol. 2013 Sep;10(9):553-62. doi: 10.1038/nrgastro.2013.107. Epub 2013 Jul 2. PMID 23817321
- [Background] European Association for Study of Liver. EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. No abstract available. PMID 25911336
- [Background] Grady BP, Schinkel J, Thomas XV, Dalgard O. Hepatitis C virus reinfection following treatment among people who use drugs. Clin Infect Dis. 2013 Aug;57 Suppl 2:S105-10. doi: 10.1093/cid/cit301. PMID 23884057
- [Background] Dore GJ, Altice F, Litwin AH, Dalgard O, Gane EJ, Shibolet O, Luetkemeyer A, Nahass R, Peng CY, Conway B, Grebely J, Howe AY, Gendrano IN, Chen E, Huang HC, Dutko FJ, Nickle DC, Nguyen BY, Wahl J, Barr E, Robertson MN, Platt HL; C-EDGE CO-STAR Study Group. Elbasvir-Grazoprevir to Treat Hepatitis C Virus Infection in Persons Receiving Opioid Agonist Therapy: A Randomized Trial. Ann Intern Med. 2016 Nov 1;165(9):625-634. doi: 10.7326/M16-0816. Epub 2016 Aug 9. PMID 27537841
- [Background] Midgard H, Bjoro B, Maeland A, Konopski Z, Kileng H, Damas JK, Paulsen J, Heggelund L, Sandvei PK, Ringstad JO, Karlsen LN, Stene-Johansen K, Pettersson JH, Dorenberg DH, Dalgard O. Hepatitis C reinfection after sustained virological response. J Hepatol. 2016 May;64(5):1020-1026. doi: 10.1016/j.jhep.2016.01.001. Epub 2016 Jan 11. PMID 26780289
- [Background] Aspinall EJ, Corson S, Doyle JS, Grebely J, Hutchinson SJ, Dore GJ, Goldberg DJ, Hellard ME. Treatment of hepatitis C virus infection among people who are actively injecting drugs: a systematic review and meta-analysis. Clin Infect Dis. 2013 Aug;57 Suppl 2:S80-9. doi: 10.1093/cid/cit306. PMID 23884071
- [Background] Sperl J, Horvath G, Halota W, Ruiz-Tapiador JA, Streinu-Cercel A, Jancoriene L, Werling K, Kileng H, Koklu S, Gerstoft J, Urbanek P, Flisiak R, Leiva R, Kazenaite E, Prinzing R, Patel S, Qiu J, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Platt HL. Efficacy and safety of elbasvir/grazoprevir and sofosbuvir/pegylated interferon/ribavirin: A phase III randomized controlled trial. J Hepatol. 2016 Dec;65(6):1112-1119. doi: 10.1016/j.jhep.2016.07.050. Epub 2016 Aug 16. PMID 27542322
- [Background] Selvapatt N, Ward T, Harrison L, Lombardini J, Thursz M, McEwan P, Brown A. The cost impact of outreach testing and treatment for hepatitis C in an urban Drug Treatment Unit. Liver Int. 2017 Mar;37(3):345-353. doi: 10.1111/liv.13240. Epub 2016 Sep 17. PMID 27566283
- [Background] Kielland KB, Amundsen EJ, Dalgard O. HCV treatment uptake in people who have injected drugs - observations in a large cohort that received addiction treatment 1970-1984. Scand J Gastroenterol. 2014 Dec;49(12):1465-72. doi: 10.3109/00365521.2014.968860. Epub 2014 Oct 13. PMID 25310139
- [Background] Mravcik V, Strada L, Stolfa J, Bencko V, Groshkova T, Reimer J, Schulte B. Factors associated with uptake, adherence, and efficacy of hepatitis C treatment in people who inject drugs: a literature review. Patient Prefer Adherence. 2013 Oct 17;7:1067-75. doi: 10.2147/PPA.S49113. PMID 24204126
- [Background] Iversen J, Grebely J, Topp L, Wand H, Dore G, Maher L. Uptake of hepatitis C treatment among people who inject drugs attending Needle and Syringe Programs in Australia, 1999-2011. J Viral Hepat. 2014 Mar;21(3):198-207. doi: 10.1111/jvh.12129. Epub 2013 Jul 1. PMID 24438681
- [Background] Lindenburg CE, Lambers FA, Urbanus AT, Schinkel J, Jansen PL, Krol A, Casteelen G, van Santen G, van den Berg CH, Coutinho RA, Prins M, Weegink CJ. Hepatitis C testing and treatment among active drug users in Amsterdam: results from the DUTCH-C project. Eur J Gastroenterol Hepatol. 2011 Jan;23(1):23-31. doi: 10.1097/MEG.0b013e328340c451. PMID 21042221
- [Background] Ferenci P, Lockwood A, Mullen K, Tarter R, Weissenborn K, Blei AT. Hepatic encephalopathy--definition, nomenclature, diagnosis, and quantification: final report of the working party at the 11th World Congresses of Gastroenterology, Vienna, 1998. Hepatology. 2002 Mar;35(3):716-21. doi: 10.1053/jhep.2002.31250. PMID 11870389
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- [Background] DAMOCLES Study Group, NHS Health Technology Assessment Programme. A proposed charter for clinical trial data monitoring committees: helping them to do their job well. Lancet. 2005 Feb 19-25;365(9460):711-22. doi: 10.1016/S0140-6736(05)17965-3. PMID 15721478
- [Derived] Vold JH, Chalabianloo F, Loberg EM, Aas CF, Lim AG, Vickerman P, Johansson KA, Fadnes LT. The efficacy of integrated hepatitis C virus treatment in relieving fatigue in people who inject drugs: a randomized controlled trial. Subst Abuse Treat Prev Policy. 2023 Apr 24;18(1):25. doi: 10.1186/s13011-023-00534-1. PMID 37095561
- [Derived] Fadnes LT, Aas CF, Vold JH, Leiva RA, Ohldieck C, Chalabianloo F, Skurtveit S, Lygren OJ, Dalgard O, Vickerman P, Midgard H, Loberg EM, Johansson KA; INTRO-HCV Study Group. Integrated treatment of hepatitis C virus infection among people who inject drugs: A multicenter randomized controlled trial (INTRO-HCV). PLoS Med. 2021 Jun 1;18(6):e1003653. doi: 10.1371/journal.pmed.1003653. eCollection 2021 Jun. PMID 34061883
- [Derived] Fadnes LT, Aas CF, Vold JH, Ohldieck C, Leiva RA, Chalabianloo F, Skurtveit S, Lygren OJ, Dalgard O, Vickerman P, Midgard H, Loberg EM, Johansson KA; INTRO-HCV Study Group. Integrated treatment of hepatitis C virus infection among people who inject drugs: study protocol for a randomised controlled trial (INTRO-HCV). BMC Infect Dis. 2019 Nov 8;19(1):943. doi: 10.1186/s12879-019-4598-7. PMID 31703669
- See also: Project web page (in Norwegian) — https://helse-bergen.no/bar